CLINICAL TRIAL: NCT05903378
Title: Early Mobilisation and Relational Touch Practice on Intubated Patients of Intensive Care Unit
Acronym: TORE-BDL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: GIRCI IDF (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP230119; 2023-A00328-37 (Other: IDRCB)
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Ventilation Therapy
Keywords: Ventilation Therapy; ICU; relational touch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relational touch group (Experimental): Touch in care aims to improve the patient's perception of potentially painful or anxiety-provoking acts of care. It is based on techniques of skin contact, developing and deepening.
  Interventions: Other: Relational touch practice
- Standard care group (No Intervention): Routine care without relational touch practice.

INTERVENTIONS:
Other: Relational touch practice — Relational touch practice during the first bedside session. Touch in care aims to improve the patient's perception of potentially painful or anxiety-provoking acts of care. It is based on techniques of skin contact, developing and deepening.
  Arms: Relational touch group

SUMMARY:
41.3% of patients hospitalized in intensive care express feeling anxiety when they are systematically questioned. Ventilatory weaning is one of the moments of anxiety for the patient. While being conscious he must tolerate invasive ventilation. The early mobilization of patients in intensive care must be started early, within 24-48 hours, after the patient wakes up. Early mobilization is part of the weaning process from invasive mechanical ventilation in intensive care. It is recommended to reduce it to use relaxation therapies. Several studies have assessed the impact of relational touch in conscious or unconscious patients in intensive care. The SRLF consensus conference in 2010 recommends the use of massage for anxiolytic purposes.

This study aims to assess the impact of relational touch versus standard care on anxiety during the first bedside session, in intubated intensive care patients ventilated for at least 48 hours and presenting with RASS (Richmond agitation sedation scale). ) from 0 to -1.

The study will aussi assess the impact of relational touch versus standard care on the following patient parameters:

* Evaluation of caregiver anxiety with the Spielberger inventory before and after the session
* Increasing the duration of the bedside session;
* Variations in pain, assessed by the Behavioral Pain Scale (BPS) at the end of the session;
* The level of agitation/vigilance at the beginning and at the end of the session with the Richmond agitation-sedation scale (RASS);
* Induced variations in blood pressure;
* Induced variations in oxygen saturation;
* The variations induced on the respiratory rate;
* The variations induced on the heart rate;
* The need to prescribe psychotropic drugs on the day of the first bedside;
* Reduction in the number of days of invasive mechanical ventilation between the first bedside session and discharge from intensive care unit (maximum D28 after the first bedside session).

This is a national, multicenter, cluster, randomized, controlled trial with 4-stage stepped-wedge design (1:1:1:1 randomization), phase III, superiority, open-label, comparing systematic practice relational touch by the paramedical team during bedside sessions, versus standard care (without relational touch).

The benefit is above all for the patient with a better experience of bedside sessions and a reduction in ventilation time, therefore bed rest, leading to a reduction in decubitus complications. The expected economic benefit involves the reduction of decubitus complications and therefore their cost and the reduction of hospitalization times in intensive care.

DETAILED DESCRIPTION:
Patient hospitalized in intensive care unit and under invasive mechanical ventilation are recruited in this research. Survivors of critical illness who are hospitalized in intensive care and have been intubated and sedated, experience a lot of problems that begin in the intensive care unit (ICU) and can continue after discharge from intensive care or even hospital.

When questioned, 41.3% of patients hospitalized in intensive care express having felt anxiety. Life in intensive care is a source of numerous, repetitive and frequent psychic traumas whose affective disorders (anxiety, stress, despair) are insufficiently detected. Barriers to better living exist in intensive care; they can be responsible for psychological manifestations such as anxiety.

One of the most distressing psychological experiences for patients receiving mechanical ventilatory support would be anxiety, defined as a state characterized by apprehension, agitation, increased motor tension, autonomic arousal and restlessness. fearful withdrawal.

Prolonged bed rest also has repercussions on the psyche of the patient who is easily anxious, confused and depressed. This prolongs the length of hospital stay. Anxiety is a feeling of dread, fear of lack of control which can manifest as agitation and fearful withdrawal, a reaction to perceived danger; also, a manifestation that can affect the psyche and physiological stability.

According to Nelson et al, between 55 and 75% of patients hospitalized in intensive care report an experience of pain, discomfort or anxiety.

At the same time, disorders of external origin (medical devices, iatrogenics) can have long-term repercussions. They can be induced by the ventilation device and result in lesions in the larynx, vocal cords, trachea such as edema, necrosis related to the balloon and pneumopathy acquired under mechanical ventilation. The objective is therefore to reduce the time of invasive ventilation in order to reduce the risk of the appearance of these complications.

Complications of a stay in intensive care or resuscitation can also be the consequence of prolonged bed rest and result in muscle weakness, cognitive disorders, psychological difficulties, reduced physical function and reduced quality of life. Early interventions such as mobilizations or active exercise, or both, can decrease the impact of severe disease sequelae. These mobilizations and this phase of ventilatory weaning themselves generate anxiety through the actions that this requires: sensory and motor stimulation, mobilization in an environment that the patient does not yet know because of his recent awakening, gestures imposed and not free due to the equipment (probes, catheters, multiple infusion lines), difficulty in expressing oneself due to the intubation probe.

Communication is the only way to prevent and try to reduce these painful experiences. Verbal and non-verbal communication (look, touch) and a body care approach are advised.

Weaning therefore generates anxiety. To reduce it, it is recommended to use relaxation therapies.

RELATIONAL TOUCH The practice of touch is part of the proper role of nurses (IDE) and caregivers (AS). It is present in more than 85% of the care provided by nurses, nursing auxiliaries and childcare auxiliaries.

Touch in care aims to improve the patient's perception of potentially painful or anxiety-provoking acts of care. It is based on techniques of skin contact, developing and deepening. It is mutually consented, intentional care. Its purpose is to communicate, reassure and provide comfort and confidence. A relational approach to create a link between the caregiver and the person cared for. Anxiolytic massages can be used in intensive care. Several studies have assessed the impact of relational touch in conscious or unconscious patients in intensive care. They demonstrate that relational touch brings relaxation and appeasement. In 47.5% of patients, a decrease in the Behavioral Pain Scale (BPS) was observed. The SRLF consensus conference in 2010 recommends the use of massage for anxiolytic purposes.

THE EDGE OF THE BED After 7 days of mechanical ventilation, 25-33% of patients have clinically evident neuromuscular weakness.

Sitting is a mobilization technique which, depending on the patient's autonomy, can be considered active, active assisted or passive active. The edge of the bed is a positioning of the patient on the edge of the bed in order to assess the patient's tolerance and capacity in the sitting position. Seated balance work can be done in bed or in an armchair. Consideration should be given to placing the patient in a seated position (bed-armchair or armchair) early on as soon as sufficient vigilance and participation have been obtained. Maintaining the seated position can be passive or active. The edge of the bed does not cause any deleterious effects for patients. Mobilization, considered as a common care by caregivers, is a source of suffering by patients described as Horror in patient testimonials.

Early mobilization involves moving the patient quickly to reduce the risks outlined above.

ACTIVE AND PASSIVE MOBILIZATION Mobilization according to its etymology from the Latin "mobilis", that is to say mobile, means that one can move, which can move easily. In the medical context mobilization is the action of moving a limb or a joint or the whole body in a passive or active way (especially after prolonged immobilization either using massage, cycling or other means exerted by the physiotherapist or by the carer on medical prescription). It is part of the process of weaning from invasive mechanical ventilation in intensive care. It must be started within 24-48 hours, following the patient's awakening and makes it possible to reduce the length of stay in intensive care. Early active mobilization makes it possible to anticipate or reduce the harmful effects of bed rest. It is as justified as passive mobilization. The implementation of passive or active mobilization is recommended as soon as possible so that the patient recovers his mobility and his autonomy in order to avoid sequelae.

BED AND ITS EFFECTS Bed rest or acute inactivity associated with hospitalization or the patient's medical condition poses a deleterious threat to functional capacity and muscle tissue.

From 24 hours of immobility, this position can have negative consequences on many functions, as described in the research of Dr. Truong:

* At the respiratory level: atelectasis, pneumonia, reduction in forced vital capacity (FVC) and reduction in maximum inspiratory pressure.
* At the cardiovascular level: decrease in the size of the heart and left ventricle, decrease in cardiac output, decrease in ejection volume, orthostatic hypotension, decrease in peripheral venous capital and function disorders circulatory.
* At the metabolic level: significant changes and disruption of endocrine activity.
* At the gastrointestinal level: disruption of transit (ileus are frequent), of the urinary system and a reduction in daily caloric intake.
* At the cutaneous level: the skin becomes fragile, which increases the risk of bedsores.
* At the musculoskeletal level: reduced muscle mass causes a decrease in strength, elasticity (connective tissues) and a loss of joint mobility (eg capsulitis) which can cause muscle atrophy.
* At the nervous level: risk of severe neuromyopathies Complications due to immobility in intensive care can persist after discharge from hospital.

Research assumptions We hypothesize that the practice of relational touch by the paramedical team during the first early mobilization session will bring about a decrease in anxiety, which could make it possible to increase the duration of bedside and possibly facilitate ventilatory weaning. .

If our study shows a decrease in anxiety in patients who have benefited from a bedside session with relational touch, the benefits will be:

* Lengthening of bed edge duration;
* Reduction in the use of psychotropic drugs;
* Reduction in the number of days of mechanical ventilation.

Benefits:

This practice will reduce stress among caregivers. Comfort care will be valued in the same way as technical care. The expected economic benefit involves the reduction of decubitus complications and therefore their cost and the reduction of hospitalization times in intensive care.

Main objective of the research To study the impact of relational touch versus standard care on patient anxiety, with the Face Anxiety Scale, during the bedside session, in intubated intensive care patients ventilated for at least 48 hours and presenting with RASS (Richmond agitation sedation scale) from 0 to -1.

Secondary objectives

To study the impact of relational touch versus standard care on the following patient parameters:

* Assessment of caregiver anxiety with the Spielberger inventory
* Increasing the duration of the bedside session
* Variations in pain, assessed by the Behavioral Pain Scale at the start and end of the session;
* The level of agitation/vigilance at the beginning and at the end of the session with the Richmond agitation-sedation scale (RASS);
* The duration of the bedside session with the scope stopwatch;
* Induced variations in blood pressure;
* Induced variations in oxygen saturation;
* The variations induced on the respiratory rate;
* The variations induced on the heart rate;
* The need to prescribe psychotropic drugs on the day of the first bedside;
* Reduction in the number of days of invasive mechanical ventilation between the first bedside session and discharge from the resuscitation and intensive care unit (maximum D28 after the first bedside session).

We will evaluate the evolution of the patient's anxiety score during the first bedside session, measured by the caregiver with the Face Anxiety Scale (FAS): difference between the beginning and the end of the bedside on the score at the Patient Anxiety Scale.

Experimental plan This is a national, multicenter, cluster, randomized, controlled trial with 4-stage stepped-wedge design (1:1:1:1 randomization), phase III, superiority, open-label, comparing systematic practice relational touch by the paramedical team during bedside sessions, versus standard care (without relational touch).

The cluster trial experimental design is indicated to avoid intervention contamination biases in this care setting (Goldstein et al., 2018); the stepped-wedge design was chosen among the types of cluster trials in view of the low risk of the intervention under study, the desire of the centers to implement this intervention eventually in their practice, to improve the power statistics and in view of the number of centers available.

Description of measures taken to reduce and avoid bias Identification of subjects

As part of this research, the subjects will be identified as follows:

center n° (3 numeric positions) - person selection order n° in the center (4 numeric positions) - surname initial - first name initial This reference is unique and will be kept for the duration of the research. Randomization The randomization of the centers (1:1:1:1) will be centralized and carried out from a list compiled in advance by the URC statistician and validated according to the procedures of the AP-HP promoter.

Randomization of centers Inclusion process (18 months) Center A Period without relational touch Formation Period with relational touch Period with relational touch Period with relational touch Period with relational touch Center B Period without relational touch Period without relational touch Formation Period with relational touch Period with relational touch Period with relational touch Center C Period without relational touch Period without relational touch Period without relational touch Formation Period with relational touch Period with relational touch Center D Period without relational touch Period without relational touch Period without relational touch Period without relational touch Formation Period with relational touch The order in which the centers will have the relational touch trainings will be decided by randomization. Each of the 5 periods will have the same start and end date (+/-15 days) for each center. For the last 4 periods, the beginning of the period will be marked by training in relational touch in one of the centers (according to the order established by randomization). The training will be carried out after the inclusion of approximately 20 patients (for 3-4 months on average, depending on the pace of recruitment) during the previous period. Inclusions will be suspended during training, but only in the center concerned by the respective training, to avoid contamination biases of the intervention under study. The centers will begin at the same time (+/- one month), with a "control" period, of inclusion of patients without relational touch (before training of caregivers). The center randomized in group A will benefit from the intervention (training of caregivers in relational touch and incentives for its use) immediately after this period (after the inclusion of approximately 20 patients for all the centers), then it will include the patients applying relational touch for all patients included and will collect data ("intervention" periods).

The centers randomized in groups B, C and D, respectively, will have respectively 2, 3 and 4 "control" periods, without application of the intervention but with information and inclusion of patients then collection of data during the bed edges carried out to these patients; then they will have training in relational touch and respectively 3, 2 and 1 periods of patient inclusion and data collection by applying relational touch for all patients ("intervention" periods; see figure above, adapted from Hooper, Bourke, BMJ 2015).

Thus, each center will have 5 patient inclusion periods (5 patients/centre/period, approximately 3 months/period) and a training phase (approximately 1-2 months) without patient inclusion. The centers should include an average of 5 patients/centre/period (between 1 and 9 patients). At the end of the study, the number of subjects with relational touch should be equal to the number of subjects without relational touch.

After the randomization of the centers, during the patient inclusion periods, all eligible patients cared for in the participating centers will be informed of this study and invited to participate by the IDEs, intensive care physicians or physiotherapists.

Eligible patients being unable to consent in writing (signing of the free and informed consent form), information on the study will be delivered to a relative of the patient present or to their trusted person if they have designated one. a. As soon as the patient is in a state to consent, he will be informed about the protocol and his agreement to continue his participation will be asked.

The edge of the bed will be carried out without a bed having a specific mechanical system but by rocking the patient in a sitting position at the edge of the bed by the 2 caregivers. Whether or not to cut the scope alarms will be decided before the start of the study with the centers (the service practices will not be modified either the services which cut the alarms continue and those which do not continue too); it will be noted if people are hard of hearing. This method will be consistent for all the centers which will use the procedures resulting from current care to carry out the mobilization of the patient.

The course of the "edge of bed" session for all the subjects will be as follows:

* The doctor prescribes the bedside session.
* The patient knows that he is participating in a study on mobilization times. After validation of the eligibility criteria and once the consent of the patient's relative or trusted person has been obtained, the first edge of the bed can be organized (with or without relational touch) according to the period of the study determined by randomization. .
* For the "intervention" periods only, caregivers are made aware of relational touch and have access to a descriptive sheet of the maneuvers.
* In the 2 or 3 caregivers (depending on the patient's tone and corpulence), the presence of at least one IDE is mandatory.
* The other carers can be another IDE, a physiotherapist or an AS.
* The ventilation mode is either controlled assisted ventilation (VAC) or spontaneous ventilation with pressure support (VSAI).
* Before entering the room, caregivers self-assess with the inventory of Spielberger Schweitzer and Paulhan
* Caregivers enter the room, inform and prepare the patient for mobilization.
* The caregivers assess the patient's anxiety with the face anxiety scale.
* The caregiver facing the scope states aloud the start time of the mobilization (T0).
* The patient is seated at the edge of the bed. Feet on the ground or not but bed height lowered to the maximum.
* One or two caregiver(s) position(s) in front of the patient to hold him (by the shoulders, hands or forearms) as well as to hold the ventilator hoses.
* Asks the patient for their self-assessment of anxiety and pain now that they are seated.

The caregiver facing the patient gives his assessment of the patient's anxiety to his colleague who collects the clinical parameters and the data related to the study in writing.

For the "intervention" periods, the carer who will practice the touch positions himself behind the patient and performs the touch maneuvers on the dorso-lumbar area, respecting the descriptive sheet. A caregiver positions himself in front of the patient to hold him and hold the ventilator hoses. The third caregiver records the parameters necessary for the clinical follow-up of the patient as well as the data related to the study. The rest of the patient care will be identical between the two groups of patients.

* The second carer records the parameters of T0, T5 and T10 (as well as T15 and T20 if applicable) (PA, SAO2, FR, FC, BPS, FAS, RASS).
* The procedure takes up to 20 minutes depending on the patient's clinical tolerance.
* For "intervention" periods only, the carer who will perform the touch (second carer) positions himself behind the patient and performs the touch maneuvers on the dorso-lumbar area, respecting the description sheet. For the "control" periods of the study, the second carer positions himself behind the patient to prevent the patient from tipping backwards but does not touch the patient if the patient is not leaning backwards.
* At the end of the session, the second carer records the TfinBDL parameters (PA, SAO2, FR, FC, BPS, FAS and RASS) and notes the start and end times of the edge of the bed.
* The patient is reinstalled in the supine position with an inclination of 30°.
* When leaving the room, caregivers self-evaluate with the inventory of Spielberger Schweitzer and Paulhan
* The IDE or AS fills in the observation notebook form, specifying the ventilation mode, the number of caregivers and their qualifications, the duration of the session and reports the parameters recorded.
* One of the caregivers who took part in the session noted the parameters (PA, SAO2, FR, HR, BPS, FAS, RASS) at TfinBDL+5.
* The IDE sends the results of the BDL test to the doctor.
* The criteria for stopping the session will be:

Heart rate < 50 or > 130/min, Systolic blood pressure < 90 mmhg or > 200 mmhg, Mean blood pressure < 60 mmhg or > 120 mmhg, Respiratory rate greater than 35/min, A loss of 5 saturation points or a saturation <90% and the patient's wishes. (Médrinal, 2012) neuro-state monitoring

• The patient's consent to continue will be requested from the patient as soon as they are able to consent, that is, after extubation and muscle recovery.

The number of days of invasive mechanical ventilation between the first bedside session and discharge from the resuscitation and intensive care unit (maximum D28 after the first bedside session) will be collected from the medical file.

Persons whose consent is sought Who informs and collects the consent of the person When the person is informed When the consent of the person is collected

* The person who agrees to the research;
* Trusted person IDEs, resuscitators or trained physiotherapists 15 min Before the treatment After a reflection period of 15 minutes at the latest when implementing a specific research procedure

Description of population

The description of the population will be made globally and by type of period: "control" and "intervention". Quantitative data will be described by their central position (mean, median) and dispersion (standard deviation, interquartile range, range) parameters and compared between patients with and without intervention using Student's or Wilcoxon's tests. Qualitative and ordinal data will be described by their frequency distribution (proportions and 95% confidence intervals) and compared between patients with and without intervention using Chi-square or Fisher tests.

Main analysis

The impact of relational touch on the evolution of the FAS score during the edge of the bed will be evaluated using a multi-level linear regression model with random effects, taking into account the variable on the intervention (patient with or without relational touch), the inclusion period (5 periods) as fixed effects and a random effect for the center.

Secondary analyzes

The impact of relational touch on the various quantitative secondary endpoints (caregiver anxiety score, BPS and RASS scores, blood pressure, oxygen saturation; respiratory rate, heart rate, psychotropic treatment duration and dosage) will be assessed. by models similar to the one used for the primary endpoint: multi-level linear regression models with random effects, taking into account the intervention variable (patient with or without relational touch), the inclusion period (5 periods) as fixed effects and a random effect for the center.

The impact of relational touch on the number of days without invasive mechanical ventilation from inclusion to discharge from the resuscitation/intensive care unit (maximum D28 after the first bedside session) will be evaluated by a Poisson regression model multi-level random effects, taking into account the intervention variable (patient with or without relational touch), the inclusion period (5 periods) as fixed effects and a random effect for the centre.

The models to meet the primary and secondary objectives will be adjusted secondarily on the comorbidities and sociodemographic characteristics of the patients and the characteristics of the centers, if the distribution of these variables proves to be unbalanced between patients with and without relational touch.

A sensitivity analysis will be carried out in secondary for the main analysis, by constructing from the main judgment criterion an ordinal variable with 3 classes with the modalities: improvement, stability and worsening of the FAS score provided by the patient. The impact of relational touch on this variable will be evaluated by a multilevel ordinal regression model with random effects, taking into account the intervention variable (patient with or without relational touch), the inclusion period (5 periods ) as fixed effects and a random effect for the center.

For parameters with at least 3 measurements during the bedside session, their evolution during the session will be modeled and plotted graphically using repeated data mixed models (with a random effect for time (T0, T5 min, T10min, T15min, T20 min, Tfin Bedside, TfinBDL+5 min) and compared between patients with and without bedside using multilevel random effects models, taking into account the intervention variable (patient with or without relational touch), the inclusion period (5 periods) as fixed effects and random effects for the center and for the time during the session.

A sensitivity analysis on the analysis of the primary judgment criterion will be carried out, to evaluate the impact of relational touch on the evolution of the FAS score during the edge of the bed treated as an ordinal variable, using a model multilevel ordinal logistic regression with random effects, taking into account the intervention variable (patient with or without relational touch), the inclusion period (5 periods) as fixed effects and a random effect for the center.

A modified intention-to-treat analysis (without imputation) will be performed on all subjects included according to the strategy prescribed for randomisation.

Given the expected low rate of missing data (<5%), no data will be imputed. The statistical analysis will be carried out at the end of the follow-up period for all patients and after the database has been frozen, according to a statistical analysis plan drawn up and validated before the basic freeze. All confidence intervals will be calculated at the first type risk of 5% bilateral and the results of the statistical tests for the analysis of the primary endpoint will be given at the threshold of 5% bilateral. Analyzes will be performed using R software (v3). They will be carried out by a biostatistician from URC Paris Saclay Ouest under the responsibility of Pr Lamiae GRIMALDI.

Rationale for sample size In the literature, the review by Thrane et al, 2019 found significant benefits of complementary therapies, including relational touch on the symptoms of patients in intensive care (including anxiety and pain). The randomized trial by Henricson et al, 2008 showed an improvement in anxiety following relational touch in patients in intensive care, without any anxiogenic care, of up to 47% of patients with improvement in the FAS score. A trial on an intervention similar to ours (music) in intensive care showed a reduction in patient anxiety (on the VAS-A score) of 19 points/100, or 36%. In our trial, we expect a clinically significant difference between patients with and without relational touch on the evolution of the FAS score during the edge of the bed, equivalent to a standard deviation.

With these assumptions (bilateral situation, alpha=0.05, power=0.8), taking into account 5% of non-evaluable patients and applying in this 4-stage stepped-wedge cluster trial an inflation factor with a coefficient intra-class correlation of 0.03 (HAS. Methodological guide Quantitative methods for evaluating interventions aimed at improving practices. June 2007), a coefficient due to the design of repeated data of 0.8 and a coefficient due to the variable size of the cluster of 0.75, corresponding to a minimum of 1 and a maximum of 9 patients/centre/period (5 patients/centre/period on average; 100 patients are needed (4 centers randomized, 25 patients/centre on average).

The completion of the observation book via the internet by the investigator thus allows the CRA to view the data quickly and remotely. The investigator is responsible for the accuracy, quality and relevance of all data entered. In addition, when they are entered, this data is immediately checked thanks to consistency checks. To this end, the investigator must validate any change in value in the CRF. These modifications are subject to an audit trail. A justification can possibly be integrated in comment.

A paper printout will be requested at the end of the study, authenticated (dated and signed) by the investigator. The original of this document will be archived by the promoter. A copy of the authenticated document must be archived by the investigator.

Management of non-conformities Any event occurring as a result of non-compliance with the protocol, the standard operating procedures, or the legislative and regulatory provisions in force by an investigator or any other person involved in the conduct of the research must be the subject of a declaration of non-compliance.These non-conformities will be managed in accordance with the promoter's procedures.

Audit The investigators undertake to accept the quality assurance audits carried out by the sponsor as well as the inspections carried out by the competent authorities. All data, all documents and reports may be subject to audits and regulations without medical secrecy being invoked.

An audit may be carried out at any time by persons appointed by the promoter and independent of the research managers. Its objective is to ensure the quality of research, the validity of its results and compliance with the law and regulations in force.

Those directing and supervising the research agree to comply with the Sponsor's requirements for an audit The audit may apply to all stages of the research, from the development of the protocol to the publication of the results and the classification of the data used or produced in the context of the research.

ELIGIBILITY:
Inclusion Criteria:

Adult patient ventilated invasively for at least 48 hours, RASS between 0 and -1 with early mobilization prescribed but not performed.

Exclusion Criteria:

* Patient needing help from another person to mobilizing
* Patient with an unstable fracture
* Patient with a recent laparotomy (less than 10 days)
* Patient under judicial protection measures
* Patient on catecholamines
* Pregnant or breastfeeding woman
* Non-communicating patient due to neuropsychiatric pathology
* Patient benefiting from a process of palliative care or moribund patient whose estimated life expectancy is less than 30 days
* Strict bed rest order
* Fraction inspired oxygen (FIO2) >50%
* Body mass index > 40 Kg/m2
* Patient having an epidural with motor impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of patients' anxiety | at baseline
  With the Face Anxiety Scale, anxiety lever of patients will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Katia Nadaud, degree of nurse, Principal Investigator — ICU, Ambroise Paré Hospital - APHP
Locations (1):
- ICU, Ambroise Paré Hospital - APHP, Boulogne-Billancourt, France